CLINICAL TRIAL: NCT03135613
Title: Kinematics of the Healthy Knee and the Surgery Knee in Patients With Tumor Around Knee After Microwave Ablation With Plate Internal Fixation.
Brief Title: Kinematics of Knees of Patients With Tumor Around Knee After Microwave Ablation With Plate Internal Fixation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Collaborators: Medical Center of Assessment, Prevention and Treatment of Bone & Joint Diseases, Guangdong, China (Other)
Responsible Party: Principal Investigator, Yu Zhang, chief surgeon, associate professor, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: GuangzhouGH009
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Knee Tumor; Microwave
Keywords: Knee tumor; Microwave; Gait
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: The control group was recruited from healthy subjects. The experimental group was recruited from patients with tumor around knee after microwave ablation with plate internal fixation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal (Experimental): Participants of this group are as controls.
  Interventions: Procedure: Procedure
- MF (Experimental): Participants of this group are patients with tumor around knee after microwave ablation with plate internal fixation.
  Interventions: Procedure: Procedure

INTERVENTIONS:
Procedure: Procedure — Once participants are eligible, they will undergo the experimental procedure. Before data collection, they will walk on a treadmill in barefoot for ten minutes to adapt the condition. The gait analysis system will collect the data while they walk on the treadmill in barefoot at self-selected gait speed.

SUMMARY:
The aim of this study is to investigate kinematics of knees of patients with tumor around knee after microwave ablation with plate internal fixation

ELIGIBILITY:
Inclusion Criteria:

1. age < 40.
2. Body mass index < 30.
3. For controls, no history of major injury or surgery in lower limbs; no symptoms of lower limbs; physical examination to test the lower limbs to be healthy.
4. For MF group, patients With Tumor Around Knee After Microwave Ablation With Plate Internal Fixation for 6 months or more.

Exclusion Criteria:

1. Body mass index >30.
2. For controls, injury or surgery in hip/knee/ankle.
3. For MF group, injury or surgery in hip/ankle;
4. Neuropathic disease.
5. Muscular disease.
6. Lack ability to finish the procedure physically or mentally.
7. Easy to fall.
8. Any other conditions that can influence gait parameters of the lower limbs.

Max Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-26 (Actual); Primary Completion 2017-05-20 (Estimated); Study Completion 2017-05-25 (Estimated)

PRIMARY OUTCOMES:
Knee flexion/extension angle at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee proximal/distal translation at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee flexion/extension angle. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee adduction/abduction angle. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee internal/external rotation angle. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee anterior/posterior translation. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee distal/proximal translation. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee medial/lateral translation. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Orthopedics, Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No